CLINICAL TRIAL: NCT04350333
Title: Efficacy of Digital Cognitive Behavioral Therapy for Insomnia (CBT-I) Intervention During Pregnancy in Prevention of Post-partum Depression: a Randomized Clinical Trial
Brief Title: Efficacy of Digital CBT-I Intervention During Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Rome G. Marconi (Other)
Responsible Party: Principal Investigator, Valeria Bacaro, Principal Investigator, University of Rome G. Marconi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UMarconi
Record Dates: First submitted 2020-04-06; First posted 2020-04-17 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Insomnia in Pregnancy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-I group (Experimental): Five sessions composed of: psychoeducation on sleep change during pregnancy and postpartum; sleep hygiene principles; stimulus control technique, sleep restriction technique (f this technique will be too difficult for the participants to be apply, a replacement and less disabling technique will be applied: sleep compression); psychoeducation on the child's sleep at birth and on the change in the sleep-wake cycle in the early stages of the child's life; cognitive control technique; cognitive reconstruction technique and de-catastrophization; relapses prevention.
  Interventions: Behavioral: CBT-I
- Assertive communication training (Active Comparator): Five sessions composed of: psychoeducation and explanation of the importance of emotional and cognitive factors for good sleep. Psychoeducation about the concept of assertiveness, explanation of the passive, aggressive and assertive style; explanation and exercises regarding self-esteem and positive self-image; explanation of the development of sleep of the child in the first years of life; explanation and exercises on the phase of the management of feedback and requests; conflict management; relapses prevention.
  Interventions: Behavioral: Assertive communication training

INTERVENTIONS:
Behavioral: CBT-I — Strategies and techniques of Cognitive behavioral therapy for insomnia adapted for pregnant women: stimulus control; sleep hygiene; sleep restriction; cognitive control etc.
  Arms: CBT-I group
Behavioral: Assertive communication training — Intervention based on improving assertive communication and regulating emotions.
  Arms: Assertive communication training

SUMMARY:
This randomized controlled trial aims to evaluate the efficacy of Cognitive Behavioral Therapy for Insomnia in pregnant women. Particularly, this study aim to explore the effect of this intervention in ameliorating insomnia symptoms and in preventing post-partum depression disorder. The experimental intervention is a digital CBT-I and the control intervention group is an assertive communication training. Both interventions include a screening phase and will be delivered in a digital way and will be composed of 5 sessions. Furthermore, both interventions protocol include a baseline, half time and follow up assessments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnancy
* Women that not consume nicotine or alcool
* BMI < 30
* Women who complains of insomnia or bad sleep quality

Exclusion Criteria:

* BMI> 30
* Complicated pregnancy
* Women who consume nicotine or alcool

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 114 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Depression | Follow up: 2 weeks post partum
  Depression symptomatology (Edinburgh Postnatal Depression Scale - EPDS). Scoring: < 8: depression not likely; 9-11: depression possible; 12-13:Fairly high possibility of depression; > 14 probable depression
Depression | Follow up: 3 months post partum
  Depression symptomatology (Edinburgh Postnatal Depression Scale - EPDS). Scoring: < 8: depression not likely; 9-11: depression possible; 12-13:Fairly high possibility of depression; > 14 probable depression
Depression | Follow up: 6 months post partum
  Depression symptomatology (Edinburgh Postnatal Depression Scale - EPDS). Scoring: < 8: depression not likely; 9-11: depression possible; 12-13:Fairly high possibility of depression; > 14 probable depression
Anxiety | Follow up: 2 weeks post partum
  Anxiety symptomatology (State-trait anxiety inventory - STAI-Y). Higher scores mean a worse outcome.
Anxiety | Follow up: 3 months post partum
  Anxiety symptomatology (State-trait anxiety inventory - STAI-Y). Higher scores mean a worse outcome.
Anxiety | Follow up: 6 months post partum
  Anxiety symptomatology (State-trait anxiety inventory - STAI-Y). Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Sleep pattern (sleep onset latency; total sleep time; wake after sleep onset; sleep efficiency) | Post intervention: after 5 weeks from the start of intervention
  sleep pattern derived from sleep diaries
insomnia symptoms | Post intervention: after 5 weeks from the start of intervention
  Insomnia severity index scores (ISI). Scoring: 0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe)
Emotion regulation | Post intervention: after 5 weeks from the start of intervention
  Emotion Regulation Questionnaire (ERQ) - Higher scores mean better outcome.

IPD SHARING:
Plan to Share IPD: Undecided